CLINICAL TRIAL: NCT00895466
Title: A Phase I-II Open Label Clinical Trial, Evaluating the Efficacy and Safety of Administration of the Therapeutic Vaccine PEP-223/CoVaccine HT, to Hormone Treatment naïve, Immunocompetent Subjects With T1-3, N0-1/x, M0 Prostate Cancer, Eligible for Hormone Therapy.
Brief Title: Efficacy and Safety Study of the Therapeutic Vaccine PEP223 in Prostate Cancer Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pepscan Therapeutics (Industry)
Collaborators: TFS Trial Form Support (Industry)
Responsible Party: Chief Medical Officer, Pepscan Therapeutics
Other Study IDs: PEP223-NL-0701
Record Dates: First submitted 2009-05-06; First posted 2009-05-08 (Estimated); Last update posted 2009-05-08 (Estimated); Status verified 2009-05

CONDITIONS: Prostate Cancer
Keywords: prostatic diseases; neoplasms; prostatic neoplasms; hormones; androgen antagonists; vaccines; peptide vaccines; adjuvants, immunological
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Diseases; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: PEP-223/CoVaccine HT

SUMMARY:
The purpose of this trial is to investigate whether treatment with this new drug will result in lower testosterone levels in men with prostate cancer. At the same time it will be investigated whether the drug induces side effects, and if so, which ones.

DETAILED DESCRIPTION:
Prostate cancer growth is influenced by the male hormone testosterone. Treatment with drugs that stop the production of testosterone often results in a decrease of the tumor or inhibition of its growth. This is particularly important prior to radiotherapy, since radiation can better be focused on the prostate with as a result less frequent or less severe side effects of the radiation.

Most of the drugs used to date to stop the production of testosterone have the disadvantage that initially they may cause a rise of testosterone levels before the production is effectively blocked. The new drug that will be investigated in this trial is a vaccine. The vaccine offers a different treatment modality since it interferes at a different level of the hormonal axis that drives the testosterone production; it will not cause an initial surge.

In this trial the vaccine will be administered three times, testosterone levels will be monitored for a total period of three months.

ELIGIBILITY:
Inclusion Criteria:

* pathological confirmed prostatic adenocarcinoma, clinical stage (c) cT1-3, cN0-1/x, cM0
* baseline testosterone levels of > 4 nmol/l
* baseline PSA level of > 10 microg/l
* eligible for hormone therapy
* willingness to comply with the protocol conditions and procedures
* willing and able to give informed consent

Exclusion Criteria:

* clinical evidence of distant metastases
* previous hormonal therapy administered specifically for prostatic carcinoma
* development of another invasive neoplastic disease during the previous 5 years, or concomitant presence of another invasive neoplastic disease, except basal cell carcinoma or squamous cell carcinoma of the skin
* primary or secondary immunodeficiency, including immunosuppressive disease or use of corticosteroids or other immunosuppressive medications
* concomitant administration - or administration during the 12 weeks preceding study inclusion - of immune enhancing medication or testosterone supplements
* concomitant radiotherapy for prostate cancer
* presence of bacterial prostatitis causing a PSA increase during the 8 weeks preceding study inclusion
* simultaneous participation in another clinical trial or participation in a clinical trial involving investigational drugs within 3 months before enrollment into the present study
* BMI > 30 kg/square meter
* previous serious reaction to a vaccine such as angioedema or anaphylaxis

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-12

PRIMARY OUTCOMES:
Testosterone suppression | after 12 weeks treatment as compared to baseline

SECONDARY OUTCOMES:
The time course of testosterone suppression | after 2, 4, 6, 8, 10 and 12 weeks treatment as compared to baseline
Effects on LH and FSH levels | after 2, 4, 6, 8, 10 and 12 weeks treatment as compared to baseline
Effects on PSA levels | after 2, 4, 6, 8, 10 and 12 weeks treatment as compared to baseline
Antibody response to PEP223/CoVaccine HT | after 2, 4, 6, 8, 10 and 12 weeks treatment as compared to baseline
Safety (adverse events, laboratory values, injection site reactions) | as applicable

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - UMC Groningen, Groningen
  - UMC Nijmegen, Nijmegen